CLINICAL TRIAL: NCT06882174
Title: Timing of Immunotherapy for the Modulation of Efficacy: a Pilot Study in Metastatic Non-Small Cell Lung Cancer
Brief Title: This Study is Comparing Morning vs Random Scheduling of Standard of Care Pembrolizumab Checkpoint Inhibitor Immunotherapy Infusions in Patients With Metastatic Non-small Cell Lung Cancer
Acronym: TIME-NSCLC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT-0038
Record Dates: First submitted 2025-03-12; First posted 2025-03-18 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Morning Infusion) (Experimental): The intervention in this study is scheduling of the time of pembrolizumab infusions. This group will have their infusion start times restricted to between 0800 AM and 1000 AM .
  Interventions: Drug: Scheduling of the time of pembrolizumab infusions
- Standard of Care (Active Comparator): This group will undergo randomized scheduling in which infusions are scheduled without respect to a specific time of day. The start time of each infusion that will occur during the study intervention period will be randomized into 1 of 3 time periods: 1000 AM to 1200 PM, 1201 PM to 1400 PM, and 1401 PM to 1700 PM. Randomization of scheduling in the Standard of Care Group approximates the typical ad hoc scheduling of infusion times done as standard of care, with reduction in potential for bias on the part of those involved in scheduling given the unblinded nature of the intervention. The time windows for the Standard of Care group have been chosen to allow infusions to be scheduled throughout the day without overlap with the specific scheduling window of the Morning Group, in order to simplify interpretation of clinical outcomes.
  Interventions: Drug: Scheduling of the time of pembrolizumab infusions

INTERVENTIONS:
Drug: Scheduling of the time of pembrolizumab infusions — The intervention in this study is scheduling of the time of pembrolizumab infusions.

SUMMARY:
This clinical trial is comparing morning infusions of the study drug (pembrolizumab) to random infusion scheduling for patients with non-small cell lung cancer.

Participants will be randomized to either the Intervention (Morning Group) where Infusion start times are restricted between 0800 AM and 1000 AM or to the Control (Standard of Care) group where scheduling will occur as standard of care scheduling, in which infusions are scheduled without respect to a specific time of day.

There are past studies that suggest the timing of treatment may influence immune response and outcomes. This idea is called chronotherapy. Chronotherapy explores the notion that the timing of drug administration in relation to the body's internal clock can optimize treatment effectiveness. The timing of the infusions for the morning group was therefore, chosen based on data from these past studies that looked at circadian variation in immune system function with the intent to focus on similar infusion windows.

The aim of this study is to provide confirmation that the intervention is possible to achieve and use these results to design a larger study. Circadian timing of drug administration, if effective, would represent an intervention that could improve survival outcomes at no additional cost or apparent increase in toxicity, which is truly rare in oncology.

Participants are asked to participate in the study intervention for 18 weeks (6 cycles of pembrolizumab), after which participants would continue with ad hoc scheduling as per standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologic diagnosis mNSCLC with PDL1 staining ≥ 50% on standard of care IHC testing
2. Patients must be eligible for treatment with standard-of-care pembrolizumab
3. Patients must be 18 years of age or older.
4. Patients must be capable of providing consent to enrolment and willing to comply with study, treatment and follow-up.
5. Patients with a performance status of Eastern Cooperative Oncology Group (ECOG) performance status 0-2 (Oken et al., 1982) will be eligible for enrolment
6. Women of childbearing potential (WOCBP) must have a negative serum (or urine) pregnancy test within 7 days prior to the first dose of pembrolizumab. WOCBP is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy or bilateral salpingectomy) and is not postmenopausal. Menopause is defined as 12 months of amenorrhea in a woman over age 45 years in the absence of other biological or physiological causes.
7. Patients of childbearing / reproductive potential should use adequate birth control methods, as defined by the investigator, during the study treatment period. A highly effective method of birth control is defined as those that result in low failure rate (i.e. less than 1% per year) when used consistently and correctly.

   Note: abstinence is acceptable if this is established and preferred contraception for the patient and is accepted as a local standard.
8. Absence of any condition hampering compliance with the study protocol and follow- up schedule; those conditions should be discussed with the patient before registration in the trial.
9. The following adequate organ function laboratory values must be met:

Hematological:

* Absolute neutrophil count (ANC) >1.0
* Platelet count >100
* Hemoglobin >90 mg/dL

Renal:

o Serum creatinine <3x upper limited of normal (ULN)

Hepatic:

* Total serum bilirubin <2x ULN
* AST and ALT <3x ULN

Coagulation:

o International Normalized Ratio (INR) <1.5x ULN (unless patient is receiving anticoagulant therapy and if PT or PTT is within therapeutic range of intended use of anticoagulants)

Exclusion Criteria:

1. Concurrent therapy with systemic therapy other than pembrolizumab (such as chemotherapy, targeted therapy, other checkpoint inhibitors, or hormonal therapy).
2. Treatment plan includes local therapy such as radiation or surgery.
3. Untreated symptomatic brain metastases, or previously treated brain metastases requiring corticosteroids for symptom control. Patients with untreated asymptomatic brain metastases, where all lesions are < 2cm in size with no vasogenic edema, are eligible.
4. Presence of leptomeningeal disease.
5. Known history of human immunodeficiency virus (HIV), active Hepatitis B or Hepatitis C. Testing for HIV, HBV or HCV is not mandatory for enrolment to study but may occur at the discretion of the investigator.
6. Active autoimmune disease that has required systemic treatment in past 12 months (i.e. with use of disease modifying agents, requiring >10mg prednisone or equivalent or other immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
7. Participant unwilling to agree to their treatment times being scheduled as per study protocol during the study treatment period (Cycles 1-6).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Rate of progression free survival at 18 weeks | The rate of PFS at will be analyzed at week 18
  PFS is defined as the time between the date of treatment initiation and the date of disease progression (determined utilizing RECIST 1.1 criteria) or death (whatever the cause), whichever occurs first. The rate of PFS at 18 weeks will be determined based on the number of participants who remain alive and whose disease has not progressed in each study arm at the 18 weeks imaging assessment. Comparison will be made to the baseline pretreatment computed tomography (CT) +/- magnetic resonance imaging (MRI) scans, to be completed within 6 weeks of treatment start.
Rate of deviation from scheduling intervention | Analysis of the scheduling intervention deviation rate will occur during the interim analysis (when 20 participants have completed the study intervention period), and ~90 days following completion of the 1-year follow-up period (end of study)
  Deviation from the scheduling intervention is defined as having occurred when a pembrolizumab infusion is started outside of the pre-specified time window. The deviation rate will be calculated both for all infusions for all study participants together, and for the infusions occurring for the participants in the individual study arms independently.
Dropout Rate | Analysis of the dropout rate will occur during the interim analysis (when 20 participants have completed the study intervention period), and ~90 days following completion of the 1-year follow-up period (end of study)
  Participant drop out is defined as voluntary withdrawal from the study prior to completion of study intervention period (between first pembrolizumab infusion and end-of-study visit at Week 19). The dropout rate will be calculated both for all study participants, and for the participants in the individual study arms independently.

OTHER OUTCOMES:
Progression free survival | The final analysis of PFS using the Log-Rank method will be scheduled to occur approximately 90 days following completion of the 1-year follow-up period for the final participant enrolled to study (i.e. end of study analysis).
  PFS is defined as the time between the date of treatment initiation and the date of disease progression (determined utilizing RECIST 1.1 criteria) or death (whatever the cause), whichever occurs first. For participants who remain alive and whose disease has not progressed, PFS will be censored on the date of last survival follow-up assessment at ~1 year after initiation of pembrolizumab treatment. PFS will be based on the disease assessment or date of death provided by the investigator.
Overall survival | The analysis of OS using the Log-Rank method will be scheduled to occur approximately 90 days following completion of the ~1-year follow-up period for the final participant enrolled to study (i.e. end of study analysis).
  OS is defined as the time between the date of treatment initiation and the date of death (whatever the cause)
Objective response rate at 18 weeks | Objective Response Rate will be analyzed at week 18
  Objective response rate (ORR) will be determined utilizing RECIST 1.1 criteria (Eisenhauer et al., 2009). Baseline staging diagnostic imaging will be compared to imaging at 18 weeks.
Treatment-related toxicity | The analysis of treatment-related toxicity will be scheduled to occur approximately 90 days following completion of the 1-year follow-up period for the final participant enrolled to study (ie., end-of-study analysis)
  Proportion of patients with all grade or grade 3 or higher treatment related immune-related toxicity as per Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Peripheral blood correlates of immune response | Peripheral blood will be collected prior to the initial pembrolizumab treatment, and then prior to each subsequent pembrolizumab infusion during the study intervention period (Week 1, 4, 7, 10, 13, 16, and 19)
  Analysis of peripheral blood for peripheral cytokine response and phenotyping of the peripheral immune cell repertoire.
Sensitivity analyses | Sensitivity analyses will be performed approximately 90 days following completion of the 1-year follow-up period for the final participant enrolled to study (end-of-study analysis)
  Participants in the Standard of Care randomized scheduling group will have a variable amount of their infusion occur in the morning or afternoon. A sensitivity analysis of PFS using the Log-Rank method will be performed including only those patients from the Standard of Care randomized scheduling group who have more than 25%, and more than 50% of their pembrolizumab infusions occurring after 1400 pm

IPD SHARING:
Plan to Share IPD: No